CLINICAL TRIAL: NCT05422066
Title: Frontline Selinexor(ATG-010) Plus R-CHOP Therapy for High-risk GCB-subtype Diffuse Large B-Cell Lymphoma
Brief Title: Selinexor Plus R-CHOP in High-risk GCB-subtype Diffuse Large B-Cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Li Zhiming (Other)
Collaborators: Antengene Corporation (Industry)
Responsible Party: Sponsor-Investigator, Li Zhiming, Chief physician, professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATG-010-MA-CL-DLBCL-002
Record Dates: First submitted 2022-06-13; First posted 2022-06-16 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: DLBCL Germinal Center B-Cell Type
Keywords: Selinexor; Xpovio; Newly Diagnosed; DLBCL; IPI 3-5
MeSH Terms: interventions — selinexor; Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Selinexor-R-CHOP (Experimental): Selinexor po 60mg once weekly, Rituximab iv 375 mg/sqm on day 1, Cyclophosphamide iv 750 mg/sqm on day 1, Doxorubicin iv 50 mg/sqm on day 1, Vincristine iv 0.5 mg/kg on day 1, Prednisone po 100mg on days 1-5 in a 21 days per cycle.
  Interventions: Drug: Selinexor; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone

INTERVENTIONS:
Drug: Selinexor — Selinexor (ATG-010# is a first-in-class, oral selective exportin 1 (XPO1) inhibitor (1,2). Selinexor functions by binding with and inhibiting the nuclear export protein XPO1 (also called CRM1), leading to the accumulation of tumor suppressor proteins in the cell nucleus along with inhibition of translation of oncoprotein mRNAs. Selinexor 60mg on day 1,8,15 for 21 days cycles
  Other Names: ATG-010; Xpovio
Drug: Rituximab — Induction Chemotherapy: 375mg/sqm, Intravenous administration on day 1 of each 3-week cycle until disease progression/stable disease, up to 6 cycles.
  Other Names: RiTUXimab Injection
Drug: Cyclophosphamide — Induction Chemotherapy: 750mg/m2, Intravenous administration on day 1 of each 3-week cycle until disease progression/stable disease, up to 6 cycles.
  Other Names: Cyclophosphamide Injection
Drug: Doxorubicin — Induction Chemotherapy: 70mg/m2, Intravenous administration on day 1 of each 3-week cycle until disease progression/stable disease, up to 6 cycles.
  Other Names: Doxorubicin Hydrochloride
Drug: Vincristine — Induction Chemotherapy: 1.4mg/m2 (Max: 2mg), Intravenous administration on day 1 of each 3-week cycle until disease progression/stable disease, up to 6 cycles.
  Other Names: Vincristine Injection
Drug: Prednisone — Induction Chemotherapy: 100mg, oral administration on day 1 to 5 of each 3-week cycle until disease progression/stable disease, up to 6 cycles.
  Other Names: Prednisone Oral Product

SUMMARY:
This is a phase II, multicenter, single-arm and open-label study to explore Selinexor in combination with standard of care R-CHOP in New Diagnosed high-risk GCB-subtype DLBCL (IPI 3-5). Approximately 35 patients plan to be enrolled in about 6-8 study sites of the study. And the objective is to Evaluate the safety and efficacy of XR-CHOP in High-Risk (IPI 3-5) GCB-subtype DLBCL.The enrollment period for this study is expected to be approximately 18 months. The study will end when all patients have completed 6 cycles treatment/follow-up since the initiation of the study drug, or the last patient has expired, has been lost to follow-up, or has withdrawn consent, whichever occurs first.

DETAILED DESCRIPTION:
This is a phase II, multicenter, single-arm and open-label study to explore Selinexor in combination with standard of care R-CHOP in New Diagnosed high-risk GCB-subtype DLBCL (IPI 3-5). Approximately 35 patients plan to be enrolled in about 6-8 study sites of the study.

Enrolled patients will be treated with 6 cycles of R-CHOP (Rituximab 375 mg/m2, cyclophosphamide 750 mg/m2 , doxorubicin 50 mg/m2 IV, vincristine 0.5 mg/kg on day 1, prednisone 100 mg po on days 1-5 in a 21 day cycle) and a fixed dose, 60 mg of selinexor, orally, weekly, each 3 week a cycle. Disease assessment will be made by positron emission tomography computed tomography (PET-CT) or PET- magnetic resonance imaging (MRI) scans (if CT is contraindicated) at screening (within 14 days of Cycle 1 Day 1). The PET-CT or PET-MRI scans (if CT is contraindicated) will be performed on Cycle 3 Day 1 (±1 week) and then every 8 weeks ± 1 week (i.e., Day 1 of odd numbered cycles) until disease progression is confirmed. The CT (or MRI) is allowed at alternating assessment time points (i.e., every 16 weeks, or every other scan) to replace PET if PET cannot be performed for every assessment.

Enrolled patients will be treated with 6 cycles of R-CHOP (Rituximab 375 mg/m2, Cyclophosphamide 750 mg/m2, Doxorubicin 50 mg/m2 IV, Vincristine 0.5 mg/kg on day 1, Prednisone 100 mg po on days 1-5 in a 21 day cycle) and a fixed dose, 60 mg of selinexor, orally, weekly, each 3 week a cycle. Treatment will continue for six cycles, or until intolerability, inadequate response, disease progression, consent withdrawal, or death, whichever occur first.

Two additional Rituximab doses (1 dose/21-day cycle) are permitted at cycles 7 and 8 if prespecified and considered standard of care per local practice. Investigators could prospectively give prespecified local radiotherapy consolidation after chemotherapy to treat a particular bulky disease site (at least 7 cm) or large mass. Additional prophylaxis or supportive care are recommended for better patient management.

The enrollment period for this study is expected to be approximately 18 months. The study will end when all patients have completed 6 cycles treatment/follow-up since the initiation of the study drug, or the last patient has expired, has been lost to follow-up, or has withdrawn consent, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following inclusion criteria to be eligible to enroll in this study:

  1. Willing and able to written informed consent (ICF) .
  2. Age ≥ 18 years and ≤ 75 years.
  3. Histologically confirmed Diffuse Large B-Cell Lymphoma of the germinal center B-cell(DLBCL) subtype by Hans.
  4. Patients no prior chemotherapy or radiotherapy for DLBCL, with the exception of no more than 5 days of treatment with glucocorticoids for symptom control.
  5. International Prognostic Index score of 3-5.
  6. Computed Tomography(CT)/Positron emission tomography (PET) positive measurable disease per the Lugano Classification 2014, having at least 1 node with longest diameter (LDi) greater than > 1.5cm or 1 extranodal lesion with LDi >1 cm.
  7. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2.
  8. Adequate bone marrow function at Screening(Except for underlying diseases, such as secondary hypersplenism due to bone marrow invasion or splenic invasion identified by the investigator).

     1. Absolute neutrophil count (ANC)≥1.5×109/L;
     2. Platelet count (PLT) ≥100×109/L(no platelet transfusion within 14 days prior to C1D1), or PLT≥ 75×109/L if due to lymphoma with bone marrow involvement.
     3. Hemoglobin (HB)≥85g/L(no red blood cell transfusion within 14 days prior to C1D1).
  9. Adequate hepatic and renal function:

     1. Aspartate aminotransferase (AST) or Alanine aminotransferase (ALT) ≤2.0 x upper limit of normal (ULN), or AST and ALT≤5.0 x ULN(if due to lymphoma involvement),
     2. Serum total bilirubin ≤2×ULN, or Serum total bilirubin ≤5×ULN if due to Gilbert syndrome or lymphoma involvement.
     3. Estimated creatinine clearance ≥ 30 mL/min (calculated using the formula of Cockroft-Gault).
  10. Participants of childearing potential must agree to use highly effective methods of contraception during the duration of the study and following the last dose of study treatment, female and male participants should continue contraception for 14 and 11 months, respectively.

      1. Female participants of childbearing potential must have a negative serum pregnancy test at screening(Non-Childbearing potential: Age >50 years and naturally amenorrhoeic for >1 year, or previous bilateral salpingo-oophorectomy, or hysterectomy).
      2. Male participants must agree to avoid sperm donation during the duration of the study and 14 months following the last dose of study treatment.

Exclusion Criteria:

* Inclusion/Exclusion Criteria:

Inclusion Criteria:

Patients must meet all of the following inclusion criteria to be eligible to enroll in this study:

1. Willing and able to written informed consent (ICF) .
2. Age ≥ 18 years and ≤ 75 years.
3. Histologically confirmed Diffuse Large B-Cell Lymphoma of the germinal center B-cell(DLBCL) subtype by Hans.
4. Patients no prior chemotherapy or radiotherapy for DLBCL, with the exception of no more than 5 days of treatment with glucocorticoids for symptom control.
5. International Prognostic Index score of 3-5.
6. Computed Tomography(CT)/Positron emission tomography (PET) positive measurable disease per the Lugano Classification 2014, having at least 1 node with longest diameter (LDi) greater than > 1.5cm or 1 extranodal lesion with LDi >1 cm.
7. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2.
8. Adequate bone marrow function at Screening(Except for underlying diseases, such as secondary hypersplenism due to bone marrow invasion or splenic invasion identified by the investigator).

   1. Absolute neutrophil count (ANC)≥1.5×109/L;
   2. Platelet count (PLT) ≥100×109/L(no platelet transfusion within 14 days prior to C1D1), or PLT≥ 75×109/L if due to lymphoma with bone marrow involvement.
   3. Hemoglobin (HB)≥85g/L(no red blood cell transfusion within 14 days prior to C1D1).
9. Adequate hepatic and renal function:

   1. Aspartate aminotransferase (AST) or Alanine aminotransferase (ALT) ≤2.0 x upper limit of normal (ULN), or AST and ALT≤5.0 x ULN(if due to lymphoma involvement),
   2. Serum total bilirubin ≤2×ULN, or Serum total bilirubin ≤5×ULN if due to Gilbert syndrome or lymphoma involvement.
   3. Estimated creatinine clearance ≥ 30 mL/min (calculated using the formula of Cockroft-Gault).
10. Participants of childearing potential must agree to use highly effective methods of contraception during the duration of the study and following the last dose of study treatment, female and male participants should continue contraception for 14 and 11 months, respectively.

    1. Female participants of childbearing potential must have a negative serum pregnancy test at screening(Non-Childbearing potential: Age >50 years and naturally amenorrhoeic for >1 year, or previous bilateral salpingo-oophorectomy, or hysterectomy).
    2. Male participants must agree to avoid sperm donation during the duration of the study and 14 months following the last dose of study treatment.

Exclusion Criteria:

Patients who meet any of the following criteria will not be enrolled:

1. DLBCL with mucosa-associated lymphoid tissue (MALT) lymphoma; composite lymphoma (Hodgkin lymphoma + NHL); Gray zone lymphoma; DLBCL transformed from Chronic Lymphocytic Leukemia (Richter Syndrome); Primary mediastinal large B-cell lymphoma (PMBCL); T-cell rich large B-cell lymphoma.
2. Known active central nervous system lymphoma or meningeal involvement at screening. Participants with a history of CNS disease treated into remission may be enrolled. The DLBCL of Testis involvement or more than two extranodal involvement.
3. Previous treatment with selinexor or other XPO1 inhibitors.
4. Contraindication to any drug contained in these regimen.
5. Major surgery <14 days of C1D1, Except for disease diagnosis.
6. Any life-threatening illness, medical condition, or organ system dysfunction which, in the Investigator's opinion, could compromise the participant's safety, or able to comply with the study procedures.
7. Uncontrolled (i.e., clinically unstable) infection requiring parenteral antibiotics, antivirals, or antifungals within 7 days prior to first dose of study treatment; however, prophylactic use of these agents is acceptable (including parenteral).
8. Subjects with known active Hepatitis B (HB) infection, active Hepatitis C (HCV) infection or Human Immunodeficiency Virus (HIV) positivity. Participants with active hepatitis B Virus (HBV) are eligible if antiviral therapy for hepatitis B has been given for >8 weeks and viral load is <100 international units per milliliter (IU/mL); participants with untreated hepatitis C Virus (HCV) are eligible if viral load is negative per institutional standard; participants with human immunodeficiency virus (HIV) are eligible if cluster of differentiation 4 (CD4+) T-cell counts ≥350 cells per microliter (cells/μL), viral load is negative and no history of acquired immunodeficiency syndrome (AIDS)-defining opportunistic infections in the last year.
9. Uncontrolled (i.e., clinically unstable) infection requiring parenteral antibiotics, antivirals, or antifungals within 7 days prior to first dose of study treatment; however, prophylactic use of these agents is acceptable (including parenteral).
10. Breastfeeding women or pregnant women.
11. In the opinion of the Investigator, participants who are below their ideal body weight and would be unduly impacted by changes in their weight.
12. Life expectancy of less than 6 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-07-26 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete Response Rate (CR) | up to 18 months
  Complete Remission (CR) rate at any time up of cycle 6 defined by Lugano 2014 defined response. Number of patients who achieved complete response after treatment by XR-CHOP

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | up to 18 months
  Overall Response Rate (ORR) per the Lugano Classification 2014 [ Time Frame: Cycle 1 Day 1 (each cycle consists of maximum 21 days) until a complete response (CR) or partial response (PR)
Progression Free Survival(PFS) | up to 18 months
  Duration from start of study treatment to Progressive disease(PD) or death (regardless of cause), whichever comes first.
Disease free survival(DFS) | up to 18 months
  To assess only the population with the best response to CR, Duration from patients who achieve CR or better time to first occurrence of PD or death(regardless of cause),whichever comes first.
Overall survival(OS) | up to 18 months
  Duration from start of study treatment to death (regardless of cause).
Safety/toxicity profile | From start of study drug administration up to 30 days after last dose of study treatment
  Adverse events as per CTCAE. V5.0. Number of Participants With Adverse Events (AEs) by Occurrence, Nature, and Severity [ Time

CONTACTS AND LOCATIONS:
Overall Officials: Zhiming Li, Ph.D, Principal Investigator — Sun Yat-sen University
Locations (6):
- China (6):
  - Department of Medical Oncology, Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The Affiliated People's Hospital of Ningbo University, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
All IPD results are used for publication,and can be shared with other investigators and sponsors
Supporting Information: Study Protocol
Time Frame: Study Protocol can be shared Starting 12 months after publication
Access Criteria: Study Protocol must not be shared with non-participants until after publication and must be authorized by the principal investigator and sponsors